CLINICAL TRIAL: NCT02982161
Title: A Randomized, Double-Blind, Multicenter, Placebo- and Active Comparator-Controlled Study to Evaluate Efficacy and Safety of MR308 in the Treatment of Acute Pain After Third Molar Tooth Extraction (STARDOM1).
Brief Title: Efficacy and Safety in a Randomised Acute Pain Study of MR308 (Tramadol/Celecoxib).
Acronym: STARDOM1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mundipharma Research GmbH & Co KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MR308-3501
Record Dates: First submitted 2016-11-25; First posted 2016-12-05 (Estimated); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Acute Pain
Keywords: Third Molar Tooth Extraction
MeSH Terms: conditions — Acute Pain | interventions — Tramadol; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- MR308 100 mg bid (Active Comparator): Tramadol/Celecoxib 100 mg
  Interventions: Drug: MR308
- MR308 150 mg bid (Active Comparator): Tramadol/Celecoxib 150 mg
  Interventions: Drug: MR308
- MR308 200 mg bid (Active Comparator): Tramadol/Celecoxib 200 mg
  Interventions: Drug: MR308
- Tramadol 100 mg qid (Active Comparator): Tramadol IR 100 mg
  Interventions: Drug: Tramadol
- Placebo (Placebo Comparator): Placebo to match MR308 and Tramadol IR
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MR308 — Over-encapsulated tablet, Dosing frequency: two times daily, Mode of administration: oral
  Other Names: Tramadol/Celecoxib
  Arms: MR308 100 mg bid; MR308 150 mg bid; MR308 200 mg bid
Drug: Tramadol — Over-encapsulated capsule, Dosing frequency: four times daily, Mode of administration: oral
  Other Names: Tramadol immediate release
  Arms: Tramadol 100 mg qid
Drug: Placebo — Capsule, Dosing frequency: four times daily, Mode of administration: oral
  Arms: Placebo

SUMMARY:
The MR308-3501 study is a multicenter, randomised, double-blind, parallel-group study in male and female adult subjects to demonstrate the efficacy of MR308 in the treatment of acute moderate to severe pain after the extraction of at least two third molars requiring bone removal.

DETAILED DESCRIPTION:
This is a multicenter double-blind, randomised, phase III study in male and female subjects with acute pain after third molar tooth extraction. The dental procedure must have involved extraction of at least two impacted third molars requiring bone removal. If only two impacted third molars are extracted, they must be ipsilateral and both require bone removal under local anaesthesia.

The Screening Visit (Visit 1) can take place up to 28 days before the planned third molar extractions. The randomisation visit (Visit 2) consists of three different sections, a part before the surgery, the part with the surgery and before randomisation, and a part with the randomisation and post-randomisation assessments. The visits 3 and 4, one respectively two days after the randomisation can be performed by telephone if the subject does not participate in the pharmacokinetic sampling.

The last dose of IMP should be taken by the subject about 72h after the initial dose and before the Completion/Discontinuation Visit (Visit 5) is performed.

The Adverse Event (AE) Follow-up Visit (Visit 6) is the last study visit and should not be done earlier than seven days after the subject's last dose of IMP. It can be performed by telephone.

ELIGIBILITY:
Inclusion Criteria:

1. Male/female subjects ≥ 18 years on the day of consent.
2. Willing and able to provide written informed consent for this study.
3. Subjects must have a planned elective dental procedure i.e. extraction of at least two impacted third molars (one of them must be mandibular) requiring bone removal, within 28 days after the Screening Visit. If only two impacted third molars are extracted, they must be ipsilateral and require bone removal.
4. If a female is of child-bearing potential, she must be using highly effective methods of contraception throughout the study, not breastfeeding, and have negative pregnancy tests prior to receiving IMP. A highly effective method of birth control is defined as one which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as sterilisation, implants, injectables, combined oral contraceptives, some IUDs (Intrauterine Device, hormonal), sexual abstinence or vasectomised partner).
5. Good general health as judged by Investigators on the basis of medical history and physical examination.
6. Willingness to comply with the study procedures and requirements.

Additional Inclusion Criteria after Surgery:

1. Third molar extractions completed without any immediate complication.
2. Tolerating oral fluids, no uncontrolled nausea/vomiting and ready to take oral analgesia.
3. The subject is alert and calm, spontaneously pays attention to caregiver, e.g. RASS = 0 (Sessler et al., 2002 & Ely et al., 2003).
4. Subjects with moderate or severe pain (qualifying PI-VAS score ≥ 45mm and < 70mm or ≥ 70mm) as a result of an oral surgical procedure under local anaesthesia and/or sedation*. This must be measured within a maximum of 6 hours after the end of the surgical procedure.

Exclusion Criteria:

1. Any abnormal laboratory value that is clinically significant in the opinion of Investigator that would compromise the safety of the subject in the study.
2. Any recent history of frequent nausea or vomiting, dizziness within the last 3 months regardless of etiology.
3. Subjects having any medical condition or treatment that is either a warning or contraindication as per the SmPC of tramadol (e.g. selective serotonin reuptake inhibitors (SSRIs), serotonin-norepinephrine reuptake inhibitors (SNRIs), tricyclic antidepressants, MAO inhibitors (within 14 days before taking IMP), antipsychotics, anticonvulsant and other seizure threshold-lowering medicinal products), celecoxib (e.g. increased risk of post-operative bleeding, active peptic ulceration, GI bleeding or inflammatory bowel disease) or paracetamol.
4. Known sensitivity and/or contraindication to tramadol, celecoxib, paracetamol, sulfonamides, opioids, NSAIDS, COX-2 inhibitors, or related compounds or formulation excipients as well as severe hypersensitivity reactions (e.g. anaphylactic shock, bronchospasm, angioedema) to any drugs.
5. Subjects who are known to have had inadequate pain relief from paracetamol, tramadol or celecoxib.
6. Subjects requiring any medication which is prohibited as per section prohibited medication.
7. Subjects who are in the Investigators opinion considered at increased risk of post-operative complications e.g. major dental infection/abscess.
8. Any history of drug or alcohol abuse, misuse, physical or psychological dependence, mood changes, sleep disturbance and functional capacity which have an impact on pain perception.
9. Significant neurological or psychiatric disorders including mental instability (unrelated to the pain) that could interfere with pain assessment; other pain that might impair the assessment of the nociceptive pain.
10. Any medical history of significant and/or inadequately controlled cardiovascular (uncontrolled high blood pressure, high risk of cardiovascular events, severe heart failure), pulmonary, hematologic, (including coagulopathy/bleeding disorders), neurological (e.g. subjects with epilepsy or those susceptible to seizures), liver disease (e.g. severe hepatic impairment), kidney disease (e.g. serum creatinine level greater than 1.5 times the upper limit of normal, impaired renal function in subjects taking diuretics, ACE-inhibitors, or angiotensin II antagonists), endocrine, immunologic, dermatologic painful conditions or any other conditions that may compromise the ability of the subject to participate in the study or might interfere with drug absorption, distribution, metabolism or excretion.
11. Previous randomisation in this study.
12. Subjects who participated in a clinical research study involving a new chemical entity or an experimental drug within 30 days of study entry (defined as the start of the Screening Period).
13. Subjects who were treated regularly with opioid analgesic or NSAIDs within 30 days prior to screening or who have received a long-acting NSAID within three days prior to the start of the surgery.
14. Subjects who have received any analgesic medication (e.g. NSAIDs, oral opioid preparations etc.) other than short-acting preoperative or intraoperative local anaesthetic agents within 12 hours before the start of the surgery or peri operatively until randomisation.
15. Subjects who are incapable of complying with the protocol.

Additional Exclusion Criteria after Surgery:

1. Serious complication during surgery and up to randomisation, including:

   * Post-operative primary and secondary bleed that cannot be controlled.
   * Subjects who did not had the third molar extraction completed as planned.
2. Post-operative medications or treatments that can have an analgesic effect or cause sedation or have amnesic effect are not permitted as these may interfere with the study assessments. These include use of ice packs, corticosteroids, nitrous oxide, benzodiazepines, alcohol, hypnotics, analgesics, opioids, other psychotropic medicinal products and any other analgesia except the provided study treatments
3. If in the Investigators opinion there are any factors that may confound the analysis of the study regarding efficacy and safety (e.g. a PI-VAS score greater than 90).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 818 (Actual)
Dates: Start 2016-12-28 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

PRIMARY OUTCOMES:
Efficacy of MR308 doses in the treatment of moderate to severe acute pain, based on the Sum of Pain Intensity Differences (SPID). | 0-4 hours
  The primary efficacy endpoint is the Sum of Pain Intensity Differences over 0-4 hours (SPID4). SPID4 is derived as the weighted Sum of Pain Intensity Differences (baseline pain - current pain), measured at different time points via the PI-VAS. Time between two consecutive measurements will be used for weighting. Larger values indicate larger pain relief.

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (2):
  - Medical Arts Health Research Group, Penticton
  - Mount Sinai Hospital, Toronto
- University Hospital Greifswald, Greifswald, Germany
- Semmelweis Egyetem Fogorvostudomnyi Kar, Budapest, Hungary
- Policlinico G.B. Rossi, Verona, Italy
- POLIMEDICA Centrum Badań, Profilaktyki i Leczenia Sp. z o.o. Sp. k., Zgierz, Poland
- Facultad de Odontología, Universitat de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Viscusi ER, Langford R, Morte A, Vaque A, Cebrecos J, Sust M, Gimenez-Arnau JM, de Leon-Casasola O. Safety of Co-Crystal of Tramadol-Celecoxib (CTC) in Patients with Acute Moderate-to-Severe Pain: Pooled Analysis of Three Phase 3 Randomized Trials. Pain Ther. 2024 Dec;13(6):1617-1631. doi: 10.1007/s40122-024-00655-w. Epub 2024 Sep 24. PMID 39316284
- [Derived] Langford R, Pogatzki-Zahn EM, Morte A, Sust M, Cebrecos J, Vaque A, Ortiz E, Fettiplace J, Adeyemi S, Lopez-Cedrun JL, Bescos S, Gascon N, Plata-Salaman C. Co-crystal of Tramadol-Celecoxib Versus Tramadol or Placebo for Acute Moderate-to-Severe Pain After Oral Surgery: Randomized, Double-Blind, Phase 3 Trial (STARDOM1). Adv Ther. 2024 Mar;41(3):1025-1045. doi: 10.1007/s12325-023-02744-2. Epub 2024 Jan 6. PMID 38183526